CLINICAL TRIAL: NCT07386106
Title: Examining the Effect of a Motor Intervention Program Applied to Children With Autism Spectrum Disorder on Autism-Related Symptoms, Gross Motor Skills, and Dual Task Performance
Brief Title: Motor Intervention, Motor Skills, and Dual Task in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gökçe Oktay, Assistant Professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IAU-GOKAEK
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Motor intervention; Dual-task performance; Gross motor skills; Motor skills
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study was designed as a pre-test-post-test controlled experimental trial including 28 children aged 4-6 years diagnosed with autism spectrum disorder (ASD). Participants were assigned to an experimental group (n = 14) and a control group (n = 14), with the sample size determined using G*Power analysis. Gross motor skills were assessed using the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition - Short Form (BOT-2), autism-related behaviors were evaluated with the Adapted Autism Behavior Checklist, and motor-cognitive performance was measured using a reaction time test. Assessments were conducted before and after the intervention period. The experimental group participated in a 12-week motor intervention program consisting of two 60-minute sessions per week in addition to their regular individual education, while the control group continued with their routine individual education only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Support Program (Experimental): The motor support program (MSP) consists of activities developed by the researchers based on the assessment protocols and designed to promote improvements in children's gross motor skills (such as throwing, jumping, catching, and running) while simultaneously engaging cognitive processes. The program includes dual-task activities that require children to perform motor tasks together with attention, reaction, and decision-making components.
  Interventions: Other: Motor Support Program
- Standard Education (No Motor Support) (No Intervention): Participants in the control group continued their individual education programs. However, they did not participate in any physiotherapy or motor support programs. Only pre- and post-test measurements were taken.

INTERVENTIONS:
Other: Motor Support Program — The motor support program (MSP) was implemented by the first researcher at a special education center for 12 weeks, with two sessions per week, each lasting 60 minutes. A structured and planned intervention program was developed for the first 10 weeks, while an "Activity Choice" approach was applied during the final 2 weeks of the intervention. During this phase, children were presented with various activity options derived from the activities implemented during the first 8 weeks and were encouraged to select and perform these activities. Within each session, at least three different game-based formats were used to target children's gross motor skills and dual-task (motor-cognitive) abilities. In the subsequent weeks, the intervention content was diversified by targeting different game formats.
  Arms: Motor Support Program

SUMMARY:
This study is designed to understand whether a structured movement (motor) program can help improve movement skills and daily functioning in young children with autism spectrum disorder (ASD).

The study will include children aged 4-6 years who have been diagnosed with ASD. Some children will take part in a 12-week motor intervention program in addition to their regular individual education at special education centers. This program will include movement activities twice a week, each session lasting about one hour. Other children will continue with their usual individual education only.

Before and after the 12-week period, all children will be assessed using simple and age-appropriate tools to evaluate their motor skills, ability to perform tasks that require both movement and attention at the same time, and autism-related behaviors. These assessments are commonly used in child development and do not involve any invasive procedures.

The goal of this study is to determine whether participating in a regular movement program can support motor development, coordination, and daily activity participation in children with ASD. Improving these skills at an early age may help children become more independent in daily life and enhance their overall quality of life.

The findings of this study may provide useful information for families, educators, and health care professionals and help improve movement-based practices in special education settings.

ELIGIBILITY:
Inclusion Criteria:

* Being between 4 and 6 years of age
* Having no health problems that would prevent participation in the study
* Having been diagnosed with autism according to the Health Board and Guidance and Research Center (RAM) report
* Not having previously participated in any motor-supported education programs (e.g., occupational therapy sessions)
* Having no additional diagnoses related to physical or intellectual disabilities other than autism spectrum disorder

Exclusion Criteria:

* The participant's failure to attend the training program for three consecutive sessions
* The participant's failure to fulfill the assigned responsibilities
* The participant's voluntary withdrawal from the study at any stage for any reason

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Motor Skills as Measured by the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition - Short Form (BOT-2 SF)" | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest).
  In this study, the short form of the Bruininks-Oseretsky Motor Competence Test-2 (BOT-2 SF), which was developed to assess the motor skill levels of individuals aged 4-21 years, was used. The short form used in the study consists of a total of eight subtests and 12 items. These subtests include fine motor accuracy, fine motor integration, manual agility, two-way coordination, balance, running speed and agility, hand-arm coordination and strength. The maximum score that can be obtained in the test is 50. As the total score increases, the level of motor skills increases.
Motor-Cognitive Skill Assessment Procedure | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest).
  Motor-cognitive skills were assessed using the Fitlight Trainer system. Four LED lights were positioned in front of each participant at 10 cm intervals, with placement adjusted according to the participant's height. The lights were activated in a random sequence. Participants were asked to count aloud from 1 to 10 while simultaneously turning off the illuminated lights by touching them with their foot. Task completion time was recorded via the mobile application connected to the Fitlight system and used to evaluate motor-cognitive performance.

SECONDARY OUTCOMES:
Adapted Autism Behavior Checklist (A-ABC): | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest).
  The Adapted Autism Behavior Checklist (A-ABC) is an assessment tool designed to determine the severity of autism spectrum disorder in children based on the level of support they require, in accordance with DSM-5 criteria. The scale was originally developed by Krug, Arick, and Almond in 1980 and was subsequently updated in 1993 and 2008. Total scores obtained from the scale range from 0 to 159, with scores of 68 and above indicating a "high likelihood of autistic disorder" (Eaves & Williams, 2006).
  Some items of the scale can be administered to all children, including nonverbal children, whereas additional items are evaluated for verbal children. Based on the scores obtained, the level of impairment associated with autism spectrum disorder and the degree of support required by the child can be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Esenyurt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruininks RH, & Oseretsky, B. D., 2010, Bruininks-Oseretsky Motor Yeterlilik Testi, İkinci Baskı, Kısa Form. Bloomington: Psychcorp.